CLINICAL TRIAL: NCT05451134
Title: Predictors and Outcomes of Dysglycemia in Pheochromocytoma and Paraganglioma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-06
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Pheochromocytoma; Paraganglioma; dysglycemia
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Catecholamines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with dysglycemia: Patients with dysglycemia in the included subjects with pheochromocytoma and paraganglioma
  Interventions: Other: Catecholamines
- patients without dysglycemia: Patients without dysglycemia in the included subjects with pheochromocytoma and paraganglioma
  Interventions: Other: Catecholamines

INTERVENTIONS:
Other: Catecholamines — Focus on whether catecholamine exposure is associated with dysglycemia in patients with pheochromocytoma and paraganglioma

SUMMARY:
The investigators will retrospectively analyze the clinical data of consecutive patients with pheochromocytomas and paragangliomas admitted between January 2018 and June 2020. The clinical characteristics of patients with and without dysglycemia will be compared, and whether surgery could improve the patients'dysglycemia will be also investigated.

DETAILED DESCRIPTION:
This retrospective cohort study will include all consecutive adult patients who underwent surgery for PHEOs and catecholamine-secreting PGLs from January 2018 to June 2020. Patients with recurrent PPGLs, those who required steroids after adrenalectomy, and those with inadequate clinical records were excluded. The patients' electronic medical files were reviewed. Patients with dysglycemia included those with diabetes, or impaired fasting glucose, or impaired glucose tolerance. Clinical history data such as age, sex, body mass index (BMI), the presence of preoperative symptoms, biochemical test results, and tumor characteristics, such as tumor diameters and locations were extracted and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* patients with surgical pathological diagnosis of pheochromocytomas and paragangliomas(PPGLs)

Exclusion Criteria:

* recurrent PPGLs
* patients who required steroids after adrenalectomy
* patients with inadequate clinical records were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study will include all consecutive adult patients who underwent surgery for pheochromocytomas and paragangliomas from January 2018 to June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline OGTT（oral glucose tolerance test）results to 6-12 months after surgery | Baseline, 6-12 months after surgery
  OGTT results （including fasting blood glucose in the text, blood glucose results at 2 hours after oral administration of 75g glucose）at baseline and 6-12 months after surgery will be recorded to assess the effect of surgery on dysglycemia

SECONDARY OUTCOMES:
random blood glucose results | baseline, 6-12 months after surgery
  random blood glucose results at baseline and 6-12 months after surgery will be recorded to assess the effect of surgery on dysglycemia
HbA1c | baseline, 6-12 months after surgery
  HbA1c results at baseline and 6-12 months after surgery will be recorded to assess the effect of surgery on dysglycemia
fasting blood glucose | baseline, 6-12 months after surgery
  fasting blood glucose results at baseline and 6-12 months after surgery will be recorded to assess the effect of surgery on dysglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Liang Zhou, Principal Investigator — National Center for Cardiovascular Diseases; Fuwai Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Xian-Liang Zhou, Beijing, Beijing Municipality, China